CLINICAL TRIAL: NCT05591326
Title: The Effect of Using Injectable Platelet-rich Fibrin with Microneedling Technique on Creeping Attachment
Brief Title: The Effect of Using Injectable Platelet-rich Fibrin on Root Surface Closure in Patients with Gingival Recession.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Berceste Guler (Other)
Responsible Party: Sponsor-Investigator, Berceste Guler, Associate Professor, Kutahya Health Sciences University
Organization: Kutahya Health Sciences University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-04/02
Record Dates: First submitted 2022-10-19; First posted 2022-10-24 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Gingival Recession; Gingival Recession, Localized
Keywords: i-PRF; creeping attachment; Keratinized gingival thickness; Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cases in RT1 class according to gingival recession depth (Experimental): Depth of gingival recession in mandibular anterior teeth, according to the 2017 Periodontal Classification, cases in RT1 class will be included.
  Interventions: Procedure: i-PRF application procedure

INTERVENTIONS:
Procedure: i-PRF application procedure — Local anesthesia will be applied to the area with gingival recession. Before the procedure, the venous blood taken from the patient will be centrifuged at 700 RPM for 3 minutes in glass and non-addition tubes to obtain i-PRF. i-TZF will be taken into a 2 cc injector. In 2020, Özsağır et al. Decortication, that is, microneedling, will be performed with insulin needle tips according to the protocol defined by Dr. Then the prepared i-PRF will be infected to the apical mucogingival junction of the keratinized gingival area. This process will be repeated once a month for 3 months. After the 3rd month, the horizontal and vertical gingival recession values will be evaluated and recorded at the end of 6 months and 1 year.

SUMMARY:
Gingival recession is the term used to describe the apical positioning of the marginal gingiva from the enamel-cementum junction. Platelet-rich fibrin (PRF) has been routinely used for more than 20 years to increase keratinized gingival thickness and to close gingival recessions due to the growth factors it contains. In the literature, there are studies evaluating the application of i-PRF with the microneedling technique, but there is no study evaluating the creeping attachment phenomenon and the closure percentage of gingival recession with the creeping attachment after the application of this technique. The aim of this study is to evaluate the closure rates of gingival recession and creeping attachment phenomenon after i-PRF application with microneedling technique. Systemically healthy and non-smoker patients older than 18 years of age with gingival recession in mandibular anterior teeth and keratinized gingival deficiency will be included. Before the procedure, the venous blood taken from the patient will be centrifuged at 700 RPM for 3 minutes in glass and non-addition tubes to obtain i-PRF. The prepared i-PRF will be infected to the apical mucogingival junction of the keratinized gingival area. This process will be repeated once a month for 3 months. After the 3rd month, the horizontal and vertical gingival recession values will be evaluated and recorded at the end of 6 months and 1 year.

DETAILED DESCRIPTION:
Gingival recession is the term used to describe the apical positioning of the marginal gingiva from the cemento-enamel junction. Gingival recession can cause hypersensitivity, pain, root caries, cervical erosion and/or abrasion, tooth loss, increased plaque accumulation as a result of exposure of the root surface to the oral environment, and therefore inflammation. Platelet-rich fibrin has been used routinely for more than 20 years to increase keratinized gingival thickness and close gingival recessions due to the growth factors it contains. In a study examining the effect of injectable platelet-rich fibrin (i-PRF) combined with free gingival graft (SDG) on SDG, it was shown that i-PRF has a positive effect on root surface closure. In the literature, studies to increase gingival thickness have reported that the application of i-PRF with microneedle is less invasive and i-PRF shows good results in increasing gingival thickness. The term creeping attachment is defined as the coronal positioning of the gingiva, especially after free gingival graft or connective tissue operations in the mandibular anterior region. There are various hypotheses explaining the mechanism of the creeping attachment - such as the contraction of collagen fibrils - but this issue has not been clarified yet. In some studies presented, it has been reported that the creeping attachment condition starts in the 2nd month postoperatively and can be seen even after 5 years. In the literature, there are studies evaluating the application of i-PRF with the microneedling technique, but there is no study evaluating the creeping attachment phenomenon and the closure percentage of gingival recession with the creeping attachment after the application of this technique. The aim of this study is to evaluate the closure rates of gingival recession and creeping attachment phenomenon after i-PRF application with microneedling technique. Systemically healthy non-smoker patients older than 18 years of age with gingival recession in mandibular anterior teeth and keratinized gingival deficiency will be included in the study. Systemic and dental anamnesis will be taken from the patient before the operation and clinical measurements will be recorded.

Periodontal indices and clinical measurements will be taken from the patients with gingival recession after Phase I treatment and oral hygiene training. The clinical periodontal measurements to be taken are as follows:

1. Plaque index (Löe&Silness): It is obtained by measuring with a periodontal probe from 4 regions of a tooth (mesial, distal, buccal and lingual).
2. Gingival index (Silness & Löe): It is obtained by measuring with a periodontal probe from 4 regions of a tooth (mesial, distal, buccal and lingual).
3. Attachment loss: It is the value of the distance between a tooth and the free gingiva by using a periodontal probe, based on the enamel-cementum junction.
4. Bleeding on probing index (Ainamo & Bay): In this index, probing is performed by gently walking around the pocket. As a result of probing, the evaluation is made by looking at the presence or absence of bleeding in the gingiva. A positive value is given if bleeding occurs within 10-15 seconds after probing in the mesial, distal, buccal and lingual parts of all teeth. The ratio of the bleeding area to the examined area is expressed as %.
5. Pocket depth: It is the vertical distance measured between a standard periodontal probe and the base of the periodontal sulcus and the gingival margin.
6. Keratinized gingival height: It is the distance from the free gingival margin to the mucogingival junction line.
7. Keratinized gingival thickness: It is the distance measured between the gingival surface and hard tissue with a standard periodontal probe inserted perpendicular to the keratinized gingiva.
8. Gingival recession depth: It is obtained by measuring the distance between the gingival margin in the midbuccal region and the enamel-cementum junction.
9. Gingival recession width: It is the amount of mesio-distal width of recession from the midpoint of the distance between the enamel cement junction and the gingival margin.
10. Keratinized mucosa thickness: After local anesthesia, it is measured with a periodontal probe or with the help of a spreader and rubber stopper.
11. Gingival phenotype: Visibility of the periodontal probe in the sulcus
12. Vestibular sulcus depth: It is the distance measured from the gingival margin to the base of the sulcus.

Obtaining Standardized Photographs Photographs of the region will be taken to measure the keratinized gingival width and gingival recession. The camera lens will be set perpendicular to the area when taking pictures. In order to determine the measurements in millimeters and to standardize the measurements on the photographs, 4.0 mm long rods of 1 mm thick round wire will be prepared. Photos will be taken in this way by placing it on the soft tissue close to the operation area. In order to standardize photographic images, images will be obtained with the same camera using the same standard magnification size.

Surgical Operation

Local anesthesia will be applied to the area with gingival recession. Before the procedure, the venous blood taken from the patient will be centrifuged at 700 RPM for 3 minutes in glass and non-addition tubes to obtain i-PRF. i-TZF will be taken into a 2 cc injector. In 2020, Özsağır et al. Decortication, that is, microneedling, will be performed with insulin needle tips according to the protocol defined by Dr. Then the prepared i-PRF will be infected to the apical mucogingival junction of the keratinized gingival area. This process will be repeated once a month for 3 months. After the 3rd month, the horizontal and vertical gingival recession values will be evaluated and recorded at the end of 6 months and 1 year.

Sample Selection: When the effect size was taken as 0.06 for the significance value in the G Power analysis program, it was planned to take 50 teeth for α= 0.05 and 80% power.

Statistical analysis method:

Gingival phenotypes will be divided into two groups as thin and thick. All analyzes will be done with the SPSS software program. Intra-temporal evaluations between the two groups will be evaluated using the Paired sample -T or Wilcoxon test according to the normal distribution values. According to the normal distribution of the data for intergroup comparisons, the Student-t test will be analyzed for parametric in-group evaluations and the Mann Withney U test for nonparametrics. The normal distribution of the data will be evaluated with the Kolmogorov-Smirnov test. Relationships between variables will be evaluated with Logistic Regression Analysis or Multivariate Regression Analysis.

ELIGIBILITY:
Inclusion Criteria:

* Be over 18 years old
* The patient does not have any systemic disease
* Presence of at least one tooth with gingival recession in the mandibular or maxillary anterior region
* Excessive dentin sensitivity and impaired esthetics associated with recession
* Identifiable enamel-cementum junction in the gingival recession area
* The tooth is alive and there are no irregularities, grooves, caries and restorations in the area to be treated.
* No periodontal surgical treatment in the relevant areas in the last 24 months
* Cases in RT1 class according to 2017 Periodontal Classification according to gingival recession depth

Exclusion Criteria:

* Being outside the specified age range
* Any contraindication for systematic periodontal surgery
* Presence of caries, restoration, root concavity in the area to be treated
* Patients who smoke more than 10 cigarettes per day
* Patients who use drugs that suppress the immune system or impair healing
* Patients using drugs that impair bleeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-09-06 (Actual); Primary Completion 2025-09-05 (Estimated); Study Completion 2025-12-04 (Estimated)

PRIMARY OUTCOMES:
The amount of root closure will be measured with the creeping attachment. | 1 year
  The amount of root surface closure will be measured with the Creeping attachment in the 1st year following the injectable platelet-rich fibrin application procedure with the microneedling technique.

CONTACTS AND LOCATIONS:
Overall Officials: Berceste Güler, Principal Investigator — Kütahya Health Sciences University Faculty of Dentistry
Locations (1):
- Kütahya Health Sciences University Faculty of Dentistry, Department of Periodontology, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared in case of contacting the research coordinator.
Supporting Information: Study Protocol, CSR
Time Frame: After the study is completed and published
Access Criteria: After the study is completed and published, the IPD will be shared if the research coordinator is contacted.

REFERENCES:
- [Background] Wan W, Zhong H, Wang J. Creeping attachment: A literature review. J Esthet Restor Dent. 2020 Dec;32(8):776-782. doi: 10.1111/jerd.12648. Epub 2020 Sep 8. PMID 32896991
- [Background] Ahrlund-Richter L, Wikstrom AC, Ramqvist T, Klein E. The Lyt phenotype of the T cells in an antitumor adoptive transfer differs for "parent to F1" and "parent to parent" combinations. Cell Immunol. 1984 Jul;86(2):575-82. doi: 10.1016/0008-8749(84)90416-7. PMID 6610486
- [Background] Miron RJ, Moraschini V, Del Fabbro M, Piattelli A, Fujioka-Kobayashi M, Zhang Y, Saulacic N, Schaller B, Kawase T, Cosgarea R, Jepsen S, Tuttle D, Bishara M, Canullo L, Eliezer M, Stavropoulos A, Shirakata Y, Stahli A, Gruber R, Lucaciu O, Aroca S, Deppe H, Wang HL, Sculean A. Use of platelet-rich fibrin for the treatment of gingival recessions: a systematic review and meta-analysis. Clin Oral Investig. 2020 Aug;24(8):2543-2557. doi: 10.1007/s00784-020-03400-7. Epub 2020 Jun 26. PMID 32591868